CLINICAL TRIAL: NCT02068768
Title: A Prospective, Multicenter, Open Label Clinical Study of the Safety andEfficacy of the Avenue L Interbody Spinal Fusion System Using the VerteBRIDGE Plating System and Supplemental Posterior Fixation
Brief Title: Multicenter Study of the Avenue L Interbody Spinal Fusion System Using VerteBRIDGE Plating and Posterior Fixation
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: LDR Spine USA (Industry)
Responsible Party: Sponsor
Other Study IDs: AveL100
Record Dates: First submitted 2014-02-19; First posted 2014-02-21 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Degenerative Disc Disease
Keywords: fusion; lateral interbody fusion system; lumbar spine; degenerative disc disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Operated Subjects: Subjects scheduled to receive an Avenue® L Interbody Fusion System (LDR Spine) for fusion of the lumbar spine from L2-S1
  Interventions: Device: Avenue® L Interbody Fusion System (LDR Spine)

INTERVENTIONS:
Device: Avenue® L Interbody Fusion System (LDR Spine) — PEEK, intervertebral cage for interbody fusion of the lumbar spine

SUMMARY:
The purpose of this prospective clinical study is to examine the short-term safety and efficacy of the Avenue®- L interbody Spinal Fusion System with VerteBRIDGE® plating to treat one and two level degenerative disc disease between L2 and S1 with a focus on fusion rate.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be candidates for on-label use of the Avenue L device (have degenerative disc disease, use only at one or two contiguous levels, posterior fixation must be used, autograft must be used in the interbody cage)
* Subject must be skeletally mature at the time of surgery, i.e. the subject must be at least 21 years of age at the time of surgery
* Subject should have had a minimum of 6 months of non-operative treatment prior to surgery
* The placement of the Avenue L device must be a primary surgery
* Subject must be willing to sign the consent form and be able to return for all follow up visits.

Exclusion Criteria:

* Subject must not have had prior surgery at the operative level(s)
* Subject is known to have substance or alcohol addictions
* Subject has lateral curvature of the spine (scoliosis, all types)
* Subject is a prisoner
* Subject is pregnant
* Subject has an active infection or sepsis at the time of surgery
* Subject has any neuromuscular disorder that would preclude accurate neurologic evaluations

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be drawn from the patient populations of the physicians participating in the study. The principal investigators include community physicians in private practice as well as physicians affiliated with academic institutions.
Sampling Method: Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2013-07-15 (Actual); Primary Completion 2016-03-09 (Actual); Study Completion 2016-03-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Center for Spine and Orthopedics, Thornton, Colorado
  - Orthopedic Surgery, Atlanta, Georgia
  - Jersey Shore University Medical Center, Neptune City, New Jersey
  - Southern New York Neurosurgical Group, Johnson City, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Operated Subjects
Started | 13
Completed | 6
Not Completed | 7
Not completed — Lost to Follow-up | 5
Not completed — Early Termination by Sponsor | 2

BASELINE CHARACTERISTICS:
Population: Subjects enrolled and completed surgery with implant of Avenue L device
Arm/Group | Operated Subjects
Number analyzed (Participants) | 13
Age, Continuous [Mean (Full Range); unit: Years] | 54.5 [30 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 12
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13
BMI (kg/m^2) [Mean (Full Range); unit: kg/m^2] | 31.5 [23.2 to 42.4]
Previous Lumbar Surgery [Count of Participants; unit: Participants] | 4
Surgical Level [Count of Participants; unit: Participants]
  L2-L3 | 3
  L3-L4 | 3
  L4-L5 | 6
  L2-L4 | 1

OUTCOME MEASURES:

1. Primary Outcome: Fusion Rate
Description: Number of participants with fused disc space as measured radiographically
Time Frame: 12 months after device implantation
Population: Poor enrollment led to early termination and low number of participants available for analysis. Data were available for 13 participants preoperatively, 12 at 3 months, 8 at 6 months, and 6 at 12 months. Only 3 of 6 participants reaching 12 month follow up had radiographs available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Operated Subjects
Number analyzed (Participants) | 3
Participants | 3

2. Secondary Outcome: Mean Oswestry Disability Index (ODI)
Description: The Oswestry Disability Index (ODI) is an index derived from the Oswestry Low Back Pain Questionnaire used by clinicians and researchers to quantify disability for low back pain. Each question is scored on a scale of 0-5 with the first statement being zero and indicating the least amount of disability and the last statement is scored 5 indicating most severe disability.The scores for all questions answered are summed, then multiplied by two to obtain the index (range 0 to 100). Zero is equated with no disability and 100 is the maximum disability possible.
Time Frame: preop, 3 mo, 6 mo, 12 mo post op
Population: Data were available for 13 participants preoperatively, 12 at 3 months, 8 at 6 months, and 6 at 12 months
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Operated Subjects
Number analyzed (Participants) | 13
score on a scale
  Preop | 53 [40 to 72]
  3 months: number analyzed (Participants) | 12
  3 months | 46 [20 to 57]
  6 months: number analyzed (Participants) | 8
  6 months | 45 [18 to 56]
  12 months: number analyzed (Participants) | 6
  12 months | 37 [0 to 47]

3. Secondary Outcome: Visual Analog Scale (VAS) of Back Pain
Description: The pain VAS is a continuous scale comprised of a horizontal line 10 centimeters in length, anchored by 2 verbal descriptors, one for each symptom extreme of either "no pain" or "worst imaginable pain". The pain VAS is self-completed by the respondent. The respondent is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0-100.
Time Frame: preop, 3 mo, 6 mo, 12 mo
Population: Data were available for 13 participants preoperatively, 12 at 3 months, 8 at 6 months, and 6 at 12 months
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Operated Subjects
Number analyzed (Participants) | 13
units on a scale
  Preop | 77 [37 to 100]
  3 months: number analyzed (Participants) | 12
  3 months | 42 [5 to 75]
  6 months: number analyzed (Participants) | 8
  6 months | 29 [0 to 67]
  12 months: number analyzed (Participants) | 6
  12 months | 23 [0 to 71]

ADVERSE EVENTS:
Time Frame: From time of surgery through 12 months post op
Description: All events deemed adverse in nature were reported. When available, a diagnosis was recorded versus a symptom. Events were assessed for relatedness to the device and include a brief description of treatment and outcome (ongoing or resolved)
Arm/Group | Operated Subjects
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 6/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Operated Subjects (N=13)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hernia (Musculoskeletal and connective tissue disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Insomnia (Psychiatric disorders) | 1 (1)
Ischemia (Cardiac disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Seroma (Investigations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Poor enrollment led to early termination and low number of participants available for analysis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No